CLINICAL TRIAL: NCT00767039
Title: Phase 4 Study of Curosurf (Poractant) and Survanta (Beractant) Surfactant Treatment in Very Premature Infants With Respiratory Distress Syndrome.
Brief Title: Curosurf and Survanta Treatment(CAST)of RDS in Very Premature Infants
Acronym: CAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment,changes in protocols, larger than anticipated differences
Sponsor: Alan Fujii (Other)
Collaborators: Dey LP (Unknown)
Responsible Party: Sponsor-Investigator, Alan Fujii, Principal Investigator, Boston Medical Center
Organization: Boston Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-23371
Record Dates: First submitted 2007-12-17; First posted 2008-10-06 (Estimated); Results first posted 2011-09-20 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2008-10

CONDITIONS: Prematurity; Respiratory Distress Syndrome; Patent Ductus Arteriosus
Keywords: Very Premature; RDS; Surfactant
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Ductus Arteriosus, Patent | interventions — beractant; poractant alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Surfactant (beractant, Survanta initial dose 100 mg/kg and subsequent doses 100 mg/kg phospholipids every 6-12 hours, as needed for up to 4 doses), intratracheal administration to very premature infants with RDS requiring mechanical ventilation
  Interventions: Drug: Survanta (beractant)
- 2 (Experimental): Surfactant (poractant, Curosurf initial dose 200 mg/kg and subsequent doses 100 mg/kg phospholipids every 12-24 hours as needed for up to 3 doses), intratracheal administration to very premature infants with RDS requiring mechanical ventilation
  Interventions: Drug: Curosurf (poractant)

INTERVENTIONS:
Drug: Survanta (beractant) — beractant 4.0 ml/kg/dose (100 mg phospholipid/kg/dose, intratracheal, every 6-12 hours as needed for respiratory distress syndrome for initial and subsequent doses, maximum of 4 doses)
  Other Names: Survanta
  Arms: 1
Drug: Curosurf (poractant) — poractant alfa 2.5 ml/kg/dose initial (200 mg phospholipid/kg), and 1.25 ml/kg/dose subsequent (100 mg/kg/subsequent dose), intratracheal, every 12-24 hours as needed for respiratory distress syndrome, maximum of 3 doses)
  Other Names: Curosurf
  Arms: 2

SUMMARY:
Approval of surfactant by the FDA in 1989 for the treatment of Respiratory Distress Syndrome (RDS) in premature infants greatly improved survival rates. Newer surfactants approved by the FDA were more concentrated and had a more rapid onset of action. The overall efficacy of newer surfactants appeared similar until in 2004, Ramanathan and colleagues suggested that a double dose of Curosurf improved survival in infants 25-32 weeks gestational age, compared to infants treated with Survanta, the most commonly used surfactant preparation in the United States. While the data was suggestive, it was not clear that the improvement in survival was reproducible or that Curosurf was responsible for the improved survival rates.

The purpose of this study was to investigate the role of Curosurf in improving lung function and survival rates and reducing the complications of prematurity in very premature infants < 30 weeks gestational age at birth.

DETAILED DESCRIPTION:
Specific Aims:

* To determine whether there is a sustained difference in the level of respiratory support during the first 3 days of life in extremely premature infants treated with Curosurf versus Survanta
* To determine whether Curosurf is associated with a higher incidence of hemodynamically significant PDA, compared with Survanta
* To determine whether there is a difference in the cerebral blood flow response to Curosurf versus Survanta
* To determine whether there is a difference in morbidity in very premature infants treated with Curosurf versus Survanta

We reasoned that if Curosurf was primarily responsible for improved survival rates, compared with Survanta, then there should be a sustained improvement in respiratory function in the first three days of life, when the direct pulmonary effects of the surfactant preparations would be most easily detected. It was also possible that Curosurf and Survanta could have effects on other systems that could secondarily affect long-term survival of the infant. These other organ systems would include, but not be limited to, the development of a hemodynamically significant Patent Ductus Arteriosus, Intraventricular Hemorrhage or Periventricular Leukomalacia, or Necrotizing Enterocolitis. We propose to examine how surfactant administration affected the hemodynamic precursors of these common morbidities of very premature infants.

ELIGIBILITY:
Inclusion Criteria:

* <29 6/7 and >24 0/7 weeks gestational age
* Inborn at the participating institution enrolling the patient
* FIO2 >25% and Intubated with mean airway pressure > 5 cm H20
* <8 hours age at randomization
* Signed informed consent from parent(s)

Exclusion Criteria:

* <500 g birth weight
* <24 0/7 weeks gestational age (best estimate)
* Prolonged Premature Rupture of membranes >3 weeks (21 days)
* Apgar score < 3 at 5 minutes
* Impending death anticipated within the first 3 days of life, moribund
* Severe congenital anomalies

Max Age: 8 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 52 (Actual)
Dates: Start 2005-01; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan M Fujii, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Fujii AM, Editorial. Is There Really A Clinical Difference In Surfactant Preparations? J Perinatol 2010; 30:698; doi:10,1038/jp.2010.90
- [Background] Fujii A. Editorial. Are all animal derived surfactants the same? The e-NeoResearch 2011; 1 (1); 50-51.
- [Result] Fujii AM, Carillo M. Animal-derived surfactant treatment of respiratory distress syndrome in premature neonates: a review. Drugs Today (Barc). 2009 Sep;45(9):697-709. doi: 10.1358/dot.2009.45.9.1418185. PMID 19956811
- [Result] Fujii AM, Patel SM, Allen R, Doros G, Guo CY, Testa S. Poractant alfa and beractant treatment of very premature infants with respiratory distress syndrome. J Perinatol. 2010 Oct;30(10):665-70. doi: 10.1038/jp.2010.20. Epub 2010 Mar 25. PMID 20336076
- [Result] Fujii A, Allen R, Doros G, O'Brien S. Patent ductus arteriosus hemodynamics in very premature infants treated with poractant alfa or beractant for respiratory distress syndrome. J Perinatol. 2010 Oct;30(10):671-6. doi: 10.1038/jp.2010.21. Epub 2010 Mar 25. PMID 20336077
- [Result] Fujii AM, Bailey J, Doros G, Sampat K, Sikes NC, Mason M, Kaiser JR. Cerebral Blood Flow Responses to Beractant and Poractant Administration. Journal of Neonatal-Perinatal Medicine 2009; 2:27-34

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients born between 1/2005 and 5/2008 with respiratory distress syndrome requiring mechanical ventilation, <30 weeks gestation, greater than 500 g and whose parents provided informed consent were included in the study. Infants with multiple congenital anomalies, significant congenital heart disease were excluded.
Groups:
- Beractant Arm: Surfactant (beractant, Survanta), intratracheal administration to very premature infants with RDS requiring mechanical ventilation (100 mg/kg initial and subsequent doses, up to 4 doses at 6-12 h intervals)
- Poractant Alfa Arm: Surfactant (poractant, Curosurf), intratracheal administration to very premature infants with RDS requiring mechanical ventilation (initial dose 200 mg/kg, subsequent doses 100 mg/kg, up to 3 doses)
Period: Overall Study
Arm/Group | Beractant Arm | Poractant Alfa Arm
Started | 27 (Two early deaths and 3 late deaths occurred in this group) | 25
Completed | 22 | 23
Not Completed | 5 | 2
Not completed — Death | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Beractant Arm | Poractant Alfa Arm | Total
Number analyzed (Participants) | 27 | 25 | 52
Age, Categorical [Count of Participants; unit: Participants] — The population is recruited from premature infants with Respiratory Distress Syndrome on the first day of life.
  Participants
    <=18 years | 27 | 25 | 52
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 13 | 20
  Male | 20 | 12 | 32
Region of Enrollment [Number; unit: participants]
  United States | 27 | 25 | 52
Gestational Age in weeks [Mean (Standard Deviation); unit: weeks] — All patients are enrolled on the first day of life. Therefore the mean +/- SD = 0 +/- 0 years.
  weeks | 26.7 (1.7) | 27.1 (1.6) | 26.9 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Comparison Respiratory Support (Mean Airway Pressure) for Survanta (Beractant) and Curosurf (Poractant) at 48 Hours After Surfactant Administration.
Description: Mean Airway Pressure delivered by mechanical ventilator or nasal CPAP (cm H20) at 48 hours following surfactant administration. A volume cycle ventilator strategy that allowed airway pressure to vary with changes in lung and chest wall compliance was used for mechanically ventilated infants, while inspired oxygen concentration was controlled by the clinical team.
Time Frame: 48 hours after surfactant administration
Population: Enrolled subjects surviving >/= 3 days were included in the analysis. Two subjects in the Survanta (beractant) groups died in this period and were eliminated from this portion of the analysis.
Measure: Mean (Standard Error); unit: cm H20
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 25 | 25
cm H20 | 8.6 (0.8) | 6.4 (0.4)
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Respiratory support were compared using a t-test for individual time points and Generalized Linear Model to account for correlations among repeated measures. Patient who survive >/= 3 days were included in the analysis; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Tested null hypothesis. T-test and Generalized Linear Model was used to assess respiratory support parameters (mean airway pressure and percent fraction of inspiratory oxygen x mean airway pressure)

2. Secondary Outcome: Comparison of Infants Successfully Extubated at 48 Hours for Curosurf (Poractant) and Survanta (Beractant) Groups
Description: Subjects successfully extubated and no longer needing positive pressure endotracheal mechanical ventilation at 48 hours after surfactant administration helps to explain the difference in mean airway pressure observed between groups.
Time Frame: 48 hours after surfactant administration
Population: Patients no longer needing positive pressure endotracheal mechanical ventilation were tallied to help explain the between group differences in mean airway pressure.
Measure: Number (90% Confidence Interval); unit: Participants successfully extubated
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 27 | 25
Participants successfully extubated | 6 [3 to 10] | 13 [9 to 17]
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p < 0.05, Mantel Haenszel; Risk Ratio (RR) = 0.43, 95% CI 2-sided [0.19 to 0.95]

3. Primary Outcome: Comparison of Respiratory Support (Mean Airway Pressure) for Curosurf (Poractant) and Survanta (Beractant) 72 Hours After Surfactant Administration
Description: Mean Airway Pressure delivered by mechanical ventilator or nasal CPAP (cm H20) at 72 hours following surfactant administration. A volume cycle ventilator strategy that allowed airway pressure to vary with changes in lung and chest wall compliance was used for mechanically ventilated infants, while oxygen concentration was controlled by the clinical team.
Time Frame: 72 hours after surfactant administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm H20
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 25 | 25
cm H20 | 7.9 (0.6) | 6.0 (0.7)
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Tested null hypothesis. T-test and Generalized Linear Model was used to assess respiratory support parameters (mean airway pressure and percent fraction of inspiratory oxygen x mean airway pressure); Test type: Superiority or Other; p < 0.05, t-test, 2 sided

4. Secondary Outcome: Comparison of Infants Successfully Extubated at 72 Hours for Curosurf (Poractant) and Survanta (Beractant) Groups
Description: Subjects successfully extubated and no longer needing positive pressure endotracheal mechanical ventilation at 72 hours after surfactant administration helps to explain the difference in mean airway pressure observed between groups.
Time Frame: 72 hours after surfactant administration
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: Participants successfully extubated
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 27 | 25
Participants successfully extubated | 8 [5 to 12] | 15 [11 to 19]
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p < 0.05, Mantel Haenszel; Risk Ratio (RR) = 0.49, 95% CI 2-sided [0.25 to 0.96]

5. Secondary Outcome: Comparison of Hemodynamically Significant Patent Ductus Arteriosus (PDA) in Patients Treated With Curosurf (Poractant) and Survanta (Beractant)
Description: Hemodynamically significant PDA, considered significant by the clinical team and having at least 2 objective echocardiographic signs (PDA > 1.5 mm diameter, retrograde diastolic flow in the descending aorta, and left atrial enlargement) were tallied. Hemodynamically significant PDA may increase lung water and decrease lung compliance, requiring increased mechanical ventilator support.
Time Frame: Hemodynamically significant PDA at > 2 days
Population: Patients with clinically and hemodynamically significant Patent Ductus Arteriosus, on evaluation at >3 days, were tallied
Measure: Number (90% Confidence Interval); unit: Subjects
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 25 | 25
Subjects | 19 [15 to 22] | 8 [5 to 12]
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p < 0.01, Mantel Haenszel; Risk Ratio (RR) = 2.38, 95% CI 2-sided [1.29 to 4.38]

6. Secondary Outcome: Changes in Blood Flow Through the Patent Ductus Arteriosus (PDA) Following Second Dose of Survanta (Beractant) and Poractant Alfa (Curosurf)
Description: Maximal changes in blood flow were assessed using Doppler echocardiography following the second surfactant dose of Survanta (beractant) or Curosurf (poractant alfa), to determine whether there was a direct effect of surfactant type on PDA size or pulmonary volume overload through the PDA. The hour interval following the second surfactant dose was selected for study, when the subjects were otherwise clinically stable, not needing additional stabilization procedures.
Time Frame: First hour after 2nd surfactant dose
Population: Population was limited to those subjects with PDA's who were treated with a second dose of surfactant, when the subjects were hemodynamically stable enough to yield meaning data.
Measure: Mean (Standard Error); unit: cc/min
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 9 | 7
cc/min
  Baseline PDA Flow, before surfactant (cc/min) | 138 (36) | 123 (45)
  Maximal PDA Flow, following surfactant (cc/min) | 169 (52) | 143 (35)
  Change in PDA Flow, following surfactant (cc/min) | 32 (42) | 20 (37)
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

7. Primary Outcome: Comparison Respiratory Support (Mean Airway Pressure x Percent Fraction of Inspired Oxygen) for Survanta (Beractant) and Curosurf (Poractant) at 48 Hours After Surfactant Administration.
Description: Mean Airway Pressure x Percent Fraction of Inspired Oxygen (FIO2) at 48 hours after surfactant administration, delivered by mechanical ventilator or nasal CPAP assesses the components of respiratory support primarily affecting blood oxygenation. This index combines these parameters so that a systematic difference in clinical management of mean airway pressure or FIO2 between groups is not mistaken for a drug effect.
Time Frame: 48 hours after surfactant administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm H20-Percent of O2
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 25 | 25
cm H20-Percent of O2 | 274 (35) | 170 (18)
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

8. Primary Outcome: Comparison Respiratory Support (Mean Airway Pressure x Percent Fraction of Inspired Oxygen) for Survanta (Beractant) and Curosurf (Poractant) at 72 Hours After Surfactant Administration.
Description: Mean Airway Pressure x Percent Fraction of Inspired Oxygen (FIO2) at 72 hours after surfactant administration, delivered by mechanical ventilator or nasal CPAP assesses the components of respiratory support primarily affecting blood oxygenation. This index combines these parameters so that a systematic difference in clinical management of mean airway pressure or FIO2 between groups is not mistaken for a drug effect.
Time Frame: 72 hours after surfactant administration
Population: as for outcome 1
Measure: Mean (Standard Error); unit: cm H20-Percent of O2
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 25 | 25
cm H20-Percent of O2 | 226 (29) | 140 (16)
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

9. Secondary Outcome: Change in Anterior Cerebral Artery Blood Flow Velocity Following Second Dose of Surfactant
Description: Percent change in Anterior Cerebral Artery blood flow velocity following the second dose of beractant, reflects the change in brain blood flow associated with surfactant administration. Blood flow velocity is measured by range gated Doppler ultrasound and brain blood flow changes in proportion to changes in arterial carbon dioxide levels, induced by surfactant administration. Variability in brain blood flow is associated with increased risk for intraventricular hemorrhage.
Time Frame: One hour following second surfactant dose at 12-24 hours after initial dose
Population: The population analyzed was limited to subjects that received second dose of surfactant and were clinically stable enough to allow Doppler assessment of cerebral blood flow during the first hour following surfactant administration.
Measure: Mean (Standard Error); unit: Percent change from baseline velocity
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 9 | 7
Percent change from baseline velocity
  Blood Flow Velocity, before surfactant (cm/sec) | 12.5 (1.5) | 22.4 (2.8)
  Peak Blood Flow Velocity, post surfactant (cm/sec) | 18.3 (2.4) | 20.4 (2.1)
  Peak Change in Blood Flow Velocity (cm/sec) | 5.6 (1.3) | -2.0 (3.1)
  Percent Change in Blood Flow Velocity (%) | 47.4 (11.9) | -1.8 (14.6)
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p < 0.01, t-test, 2 sided

10. Secondary Outcome: Patients With Bronchopulmonary Dysplasia (Supplemental Oxygen at 36 Week Post Menstrual Age)
Description: Patients with Bronchopulmonary Dysplasia (BPD), had chronic lung disease requiring supplemental oxygen support at >/= 36 weeks post menstrual age, were tallied. BPD is a chronic lung disease that develops, at least in part, as a consequence of NICU respiratory management of premature infants with Respiratory Distress Syndrome.
Time Frame: 36 weeks post menstrual age
Population: Population analyzed was limited to those subjects who survived to >36 weeks post menstrual age. Subjects with Bronchopulmonary Dysplasia (continuous supplemental oxygen need at >36 weeks post menstrual age) were tallied.
Measure: Number (90% Confidence Interval); unit: Surviving Subjects with BPD
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 22 | 23
Surviving Subjects with BPD | 11 [7 to 15] | 8 [4 to 11]
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p > 0.05, Mantel Haenszel; Risk Ratio (RR) = 1.44, 95% CI 2-sided [0.71 to 2.89]

11. Secondary Outcome: Bronchopulmonary Dysplasia (Supplemental Oxygen at 36 Week Post Menstrual Age) or Death Before Discharge From NICU.
Description: Bronchopulmonary Dysplasia + death outcome for all patients enrolled in the study were tallied and used to determine whether neonatal death decreased the frequency of chronic lung disease in one group vs the other.
Time Frame: NICU hospitalization, up to 42 weeks post menstrual age
Population: All subjects enrolled were included. Subjects with Bronchopulmonary Dysplasia (continuous supplemental oxygen need at > 36 weeks post menstrual age) and patients who expired before discharge from the NICU were tallied.
Measure: Number (90% Confidence Interval); unit: Subjects with BPD + Neonatal Deaths
Arm/Group | Beractant Arm | Poractant Alfa Arm
Number analyzed (Participants) | 27 | 25
Subjects with BPD + Neonatal Deaths | 16 [12 to 20] | 10 [6 to 14]
Statistical Analysis 1: Comparison: Beractant Arm vs Poractant Alfa Arm; Test type: Superiority or Other; p > 0.05, Mantel Haenszel; Risk Ratio (RR) = 1.48, 90% CI 2-sided [0.84 to 2.63]

ADVERSE EVENTS:
Time Frame: Adverse events occurring during the NICU admission, up to 42 weeks post menstrual age.
Description: Severe adverse evens include: severe intraventricular hemorrhage, severe pulmonary hemorrhage, Necrotizing enterocolitis, Threshold Retinopathy of prematurity requiring Laser therapy, or death
Arm/Group | Beractant Arm | Poractant Alfa Arm
Serious Adverse Events (participants affected / at risk) | 19/27 | 9/25
Other Adverse Events (participants affected / at risk) | 17/27 | 8/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Beractant Arm (N=27) | Poractant Alfa Arm (N=25)
Death (General disorders) | 5 (5) | 2 (2) — Death before NICU discharge
Necrotizing Enterocolitis (Gastrointestinal disorders) | 4 (4) | 4 (4) — Stage 2 Necrotizing enterocolitis
Severe Intraventricular Hemorrahge (Grade 3-4) (Nervous system disorders) | 1 (1) | 1 (1)
Significant Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) — Pulmonary hemorrhage associated with an increase in respiratory support
ROP Stage II-IV (Eye disorders) | 10/23 (10) | 7/24 (7) — Retinopathy of Prematurity at threshold, treated with Laser
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Beractant Arm (N=27) | Poractant Alfa Arm (N=25)
Bronchopulmonary Dysplasia (Respiratory, thoracic and mediastinal disorders) | 11/22 (11) | 8/23 (8) — Oxygen requirement at 36 weeks Post menstrual age in infants surviving to 36+ weeks.
Patent Ductus Arteriosus ligation (Cardiac disorders) | 7/25 (7) | 4 (4) — PDA requiring surgical ligation
Pulmonary Air Leak (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) — Pulmonary air leak including: pulmonary interstitial emphysema, pneumothorax, pneumatocele

LIMITATIONS AND CAVEATS:
The primary limitations are the small number of patients, the high rate of chronic lung disease in the beractant group and the open-label design of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less